CLINICAL TRIAL: NCT01833429
Title: Circadian Autonomic Disturbances in Resistant Hypertension With and Without White-coat Phenomenon
Brief Title: Autonomic Dysfunction in Resistant Hypertension
Acronym: RH
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Valéria Nasser Figueiredo, PhD, University of Campinas, Brazil
Other Study IDs: 907/2011
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Resistant hypertension; White-coat phenomenon; Heart rate variability; autonomic activity
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Resistant Hypertension: The current definition of resistant hypertension (RH) includes both patients whose blood pressure (BP) is uncontrolled on three or more medications and those whose BP is controlled when using four or more antihypertensive medications

SUMMARY:
The contribution of this study is the unedited evaluation of the circadian autonomic profiles of resistant hypertension with and without white-coat response.

DETAILED DESCRIPTION:
All patients were submitted to office blood pressure measurement, Ambulatory blood pressure monitoring and 24-hour Holter monitoring.

Baseline blood samples for the measurement of glycemia (mg/dL), total cholesterol (mg/dL), LDL cholesterol (mg/dL), triglycerides (mg/dL), creatinine (mg/dL), serum uric acid, serum sodium, serum potassium, plasma aldosterone concentration (PAC) and plasma renin activity (PRA) were collected at 08:00 after overnight fasting.

ELIGIBILITY:
Inclusion Criteria:

* resistant hypertensive patients

Exclusion Criteria:

* White-coat hypertension
* obstructive sleep apnea

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Forty-four resistant hypertension subjects, regularly followed up at the cardiovascular clinical pharmacology out-patients' clinic, and who complied with pharmacological prescription for hypertension, were recruited to participate in this transversal and observational study.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
evaluation of the autonomic function in resistant hypertensive patients | 10 months
  The autonomic nervous system can be assessed by the heart rate variability. Variations in heart rate variability are normally observed in association with diurnal rhythms and blood pressure changes. The heart rate variability parameters are different in many studies, although the consensus is that lower values of the indices of vagal as well as high indices of sympathetic functions are associated prospectively with death and disability.
  In humans, the disturbances of the circadian rhythms of heart rate variability and blood pressure have been intensively studied, mainly due to the increased cardiovascular death reported during the morning hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Pharmacology Laboratory, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Result] Muxfeldt ES, Fiszman R, de Souza F, Viegas B, Oliveira FC, Salles GF. Appropriate time interval to repeat ambulatory blood pressure monitoring in patients with white-coat resistant hypertension. Hypertension. 2012 Feb;59(2):384-9. doi: 10.1161/HYPERTENSIONAHA.111.185405. Epub 2012 Jan 3. PMID 22215711